CLINICAL TRIAL: NCT06551207
Title: Fuquinitinib Combined With Cardonilizumab and SBRT Versus Fuquinitinib in Third-line and Post-line Treatment of Metastatic Colorectal Cancer: a Randomized, Controlled, Open, Multicenter Clinical Study
Brief Title: Cadonilimab Combined With Fruquintinib and SBRT as Athird-line and Posterior Line Treatment in Patients With MSS CRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Huang (Other)
Responsible Party: Sponsor-Investigator, Liu Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024TJCR020
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fuquintinib (Placebo Comparator)
  Interventions: Drug: Fruquintinib
- Fuquintinib combined with cardonilizumab and SBRT (Experimental)
  Interventions: Drug: Fruquintinib; Drug: Cadonilimab; Radiation: SBRT

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib:5mg ,qd,po, d1-d14, q3w
Drug: Cadonilimab — Cadonilimab:10mg/kg, ivgtt, d1, q3w
  Arms: Fuquintinib combined with cardonilizumab and SBRT
Radiation: SBRT — SBRT:8-10Gy×5F, god, in 10 days
  Arms: Fuquintinib combined with cardonilizumab and SBRT

SUMMARY:
An assessment of 6-month progression-free survival in patients with mCRC with third-line and postline metastatic colorectal cancer in combination with cardonilizumab and fuquinitinib and SBRT compared with fuquinitinib monotherapy

ELIGIBILITY:
Inclusion Criteria:• Provision of written Informed Consent Form (IC) prior to any study specific procedures

* Age = 18 years, $75 years
* Histologically or cytologically confirmed advanced Stage IV primary colorectal cancer
* MSI status: MSS
* At least two or more standard systemic therapies prior treatment (based on Fu, oxaliplatin, irinotecan, bevacizumab and cetuximab) of cytotoxic chemotherapy, treatment failure or intolerable toxicities
* ECOG 0-1
* Patients must have measurable lesions
* Expected overall survival ≥ 12 weeks
* AST, ALT and alkaline phosphatase s 2.5 times the upper limit of normal (ULN), Serum bilirubin s 1.5 x ULN, creatinine<ULN
* Prothrombin time (PT), international standard ratio (INR) ≤ 1.5 × ULN
* Patients are allowed to have received radiotherapy, but the time from entering the group must be more than 4 weeks, and the currently selected radiotherapy lesions and evaluable lesions must be lesions that have not received radiotherapy
* Fertile male or female patients voluntarily used an effective contraceptive method during the study period and within 6 months of the last study medication

Exclusion Criteria:

* • Patients have received anti-PD-1 / PD-L1 or anti-CTLA-4 immunotherapy or other immunexperimental drugs

  * Patients with severe autoimmune diseases: active inflammatory bowel disease (including Cohn's disease and ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus ervthematosus, autoimmune vasculitis (such as Wegener's granuloma), etc
  * Symptomatic interstitial lung disease or active infection/non-infectious pneumonia
  * Risk factors of intestinal perforation: active diverticulitis, abdominal abscess, gastrointestinal obstruction, abdominal cancer or other known risk factors of intestinal perforation
  * If the patients underwent surgery, they should wait for the wound to heal completely before being considered for enrollment
  * History of other malignant tumors ((except for the cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, and breast carcinoma in situ)
  * Patients who are preparinq for or have previously received an organ or allogenic bone marrow transplant
  * Moderate or severe ascites with clinical symptoms required therapeutic puncture, drainage or Child-Pugh score > 2 (except those who only show a small amount of ascites on imaging without clinical symptoms); Uncontrolled or moderate or higher pleural effusion or pericardial effusion
  * History of gastrointestinal bleeding or a definite tendency to gastrointestinal bleeding within 6 months before the start of treatment
  * Abdominal fistula, gastrointestinal perforation, or abdominal abscess developed within 6 months before the start of study treatment
  * Known hereditary or acquired bleeding (e.g. coagulation dysfunction) or thrombotic tendencies, e.g. in hemophiliacs; Currently or recently (within 10 days prior to the start of study therapy) used full dose oral or injectable anticoagulants or thrombolytic agents for therapeutic purposes (allowing prophylactic use of low-dose aspirin, low molecular weight heparin)
  * Aspirin (> 325 mg / day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel (≥ 75 mg) and clostazol are currently used or have been used recently (within 10 days before the start of study treatment)
  * Thrombosis or embolism events such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction) and pulmonary embolism occurred within 6 months before the start of the study
  * Patient with an active infection, heart failure, heart attack, unstable angina pectoris, or unstable arrhythmia within the last 6 months
  * Physical examination or clinical trial findings that the investigator believes may interfere with the results or put the patient at increased risk for treatment complications, or other uncontrollable diseases
  * The researchers believe that the patient has a lesion and needs emergency palliative radiotherapy / emergency surgery (spinal cord compression, brain hernia, pathological fracture)
  * Lactating or pregnant women
  * History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation
  * Patients with mental illness, substance abuse, or social problems that affect compliance will not be enrolled after researcher's review
  * Known active infection and active tuberculosis infection were not included in the group; However, patients with hepatitis B virus (HBV) and hepatitis C virus (HCV) infection can be included in the group if their condition is stable after antiviral treatment
  * Patients who received live vaccine within 30 days prior to enrollment
  * Have clinical symptoms or diseases of the heart that are not well controlled
  * Systolic blood pressure > 140mmg or diastolic blood pressure > 90mmg regardless of any antihypertensive drugs; or a history of hypertensive crisis or hypertensive encephalopathy
  * Major vascular disease (such as aortic aneurysms requiring surgical repair or recent peripheral arterial thrombosis developed within 6 months
  * Severe, unhealed or open wounds and active ulcers or untreated fractures
  * Received major surgery within 4 weeks prior to the start of study treatment (except for diagnosis or expected to require major surgery during the study period
  * Inability to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption
  * Had a history of intestinal obstruction and/or had clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to initiation of study therapy, including incomplete obstruction related to pre-existing disease or requiring routine parenteral hydration, parenteral nutrition, or tube feeding
  * Patients with signs/symptoms of incomplete obstruction/obstructive syndrome/ileus at initial diagnosis may be admitted to the study if they have received definitive (surgical) treatment to resolve symptoms
  * There is evidence of abdominal gas accumulation that cannot be explained by puncture or recent surgical procedures
  * Metastatic disease involvina a maior airway or blood vessel or a large mediastinal tumor mass located in the center (<30 mm from the crest)
  * Patients with a history of hepatic encephalopathy For those who currentlv have interstitial oneumonia or interstitial luna disease, or who have a history of interstitial pneumonia or interstitial luna disease requiring hormone therapv. Or other
  * Patients with a history of hepatic encephalopathy
  * For those who currently have interstitial pneumonia or interstitial lung disease, or who have a history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, Or other subjects with pulmonary fibrosis, institutionalized pneumonia, pneumoconiosis, drug-related pneumonia, idiopathic pneumonia that may interfere with the judgment and management of immune-related pulmonary toxicity, or with evidence of active pneumonia or severe impairment of lung function visible on chest CT during the screening period, radiation pneumonia is allowed in the radiation field: Active tuberculosis
  * Presence of active autoimmune disease or history of autoimmune disease with possible recurrence; Participants with non-systemic skin diseases such as vitiligo, psoriasis, and alopecia, controlled type 1 diabetes treated with insulin, or asthma in complete remission in childhood, were enrolled without any intervention as adults; Patients with asthma who require medical intervention with bronchodilators are not included
  * Use of immunosuppressants or systemic hormone therapy for immunosuppression within 14 days prior to initiation of study therapy
  * Known history of severe allergy to any monoclonal antibody, anti-angiogenesis targeting drug Severe infection, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia, in the 4 weeks prior to initiation of study treatment; Therapeutic antibiotics were given orally or intravenously within 2 weeks prior to the start of study therapy
  * According to the investigator's judgment, the patient has other factors that may affect the study results or lead to the forced termination of the study. There are serious abnormalities in laboratory examination, accompanied by family or social factors, which will affect the safety of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6mon-PFS
  6-month progression-free survival in patients with third-line and postline metastatic colorectal cancer mCRC with cardonilizumab combined with fuquinitinib and SBRT compared with fuquinitinib monotherapy (6mon-PFS)

SECONDARY OUTCOMES:
Obiective response rate (ORR) | up to 42 months]
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate (DCR) | up to 42 months]
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Overall survival (OS) | up to 42 months]
  The time interval between the start date of study drug and the date of death (any cause)
quality of life (QOL) | up to 42 months]
  OOL according to OOL-C30
AEs | up to 42 months]
  Adverse reactions refer to the occurrence and development of diseases in the process of using drugs according to normal usage and dosage to prevent, diagnose or treat diseases. Adverse reactions unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No